CLINICAL TRIAL: NCT03892798
Title: Database Of Clinical Data For Individuals With Variants In The IRF2BPL Gene
Acronym: IRF2BPL
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Loren Pena, Associate Professor, Children's Hospital Medical Center, Cincinnati
Other Study IDs: 2018-6357
Record Dates: First submitted 2019-01-25; First posted 2019-03-27 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder; Movement Disorders; Seizures; Dystonia; NEDAMSS
Keywords: IRF2BPL; NEDAMSS; dystonia; movement disorder; seizures
MeSH Terms: conditions — Autism Spectrum Disorder; Movement Disorders; Seizures; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — If available left-ever tissue and blood from clinical investigations may be stored in the CCHMC Biorepository for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions are planned — No interventions are planned

SUMMARY:
This protocol serves as a data collection tool for individuals with variants (missense, nonsense, frameshifts) in the IRF2BPL gene (MIM 611720), which causes Neurodevelopmental Regression, Seizures, Autism and Developmental Delay (NEDAMSS, MIM 618088) and may be involved in other neurodevelopmental presentations. This information will be analyzed to develop a better understanding of the findings and progression of symptoms in individuals with variants in the IRF2BPL gene.

DETAILED DESCRIPTION:
Neurodevelopmental Regression, Abnormal Movements, Loss of Speech, and Seizures (NEDAMSS) is caused by changes in the IRF2BPL gene. Variants in the gene can also lead to other neurodevelopmental presentations. Due to the limited number of cases that have been described to date, clinicians may have a limited understanding of what types of symptoms can develop in affected individuals and at what age. The purpose of the study is to gather clinical information about progression, treatments and outcomes for patients with variants in IRF2BPL. The investigators will collect information about medical history, growth, development, treatments and the results of previous genetic tests. In some cases, the investigators may also collect tissue samples. This is a non-interventional study that will expand the current understanding of the range of health concerns that can be seen in individuals with changes in the IRF2BPL gene by collecting medical information and samples from a larger group of affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased individuals with variants in the IRF2BPL gene

Exclusion Criteria:

* None

Ages: 2 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of children and adults who are diagnosed with NEDAMSS and have variants in the IRF2BPL gene.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Throughout study completion, with the assessment completed on average once per year.
  The investigators will collect information regarding age at development of symptoms, age at diagnosis, method for diagnosis, specific mutations detected, additional complications with age at onset and treatment.

SECONDARY OUTCOMES:
Genotype-phenotype correlations | Throughout study completion, with the assessment completed on average once per year.
  The investigators will assess for correlations between the type of variant in the IRF2BPL gene, the location of the variant, and the clinical presentation and symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcogliese PC, Shashi V, Spillmann RC, Stong N, Rosenfeld JA, Koenig MK, Martinez-Agosto JA, Herzog M, Chen AH, Dickson PI, Lin HJ, Vera MU, Salamon N, Graham JM Jr, Ortiz D, Infante E, Steyaert W, Dermaut B, Poppe B, Chung HL, Zuo Z, Lee PT, Kanca O, Xia F, Yang Y, Smith EC, Jasien J, Kansagra S, Spiridigliozzi G, El-Dairi M, Lark R, Riley K, Koeberl DD, Golden-Grant K; Program for Undiagnosed Diseases (UD-PrOZA); Undiagnosed Diseases Network; Yamamoto S, Wangler MF, Mirzaa G, Hemelsoet D, Lee B, Nelson SF, Goldstein DB, Bellen HJ, Pena LDM. IRF2BPL Is Associated with Neurological Phenotypes. Am J Hum Genet. 2018 Sep 6;103(3):456. doi: 10.1016/j.ajhg.2018.08.010. No abstract available. PMID 30193138
- [Background] Tran Mau-Them F, Guibaud L, Duplomb L, Keren B, Lindstrom K, Marey I, Mochel F, van den Boogaard MJ, Oegema R, Nava C, Masurel A, Jouan T, Jansen FE, Au M, Chen AH, Cho M, Duffourd Y, Lozier E, Konovalov F, Sharkov A, Korostelev S, Urteaga B, Dickson P, Vera M, Martinez-Agosto JA, Begemann A, Zweier M, Schmitt-Mechelke T, Rauch A, Philippe C, van Gassen K, Nelson S, Graham JM Jr, Friedman J, Faivre L, Lin HJ, Thauvin-Robinet C, Vitobello A. De novo truncating variants in the intronless IRF2BPL are responsible for developmental epileptic encephalopathy. Genet Med. 2019 Apr;21(4):1008-1014. doi: 10.1038/s41436-018-0143-0. Epub 2018 Aug 31. PMID 30166628